CLINICAL TRIAL: NCT01677169
Title: Double Blind, Randomized, Placebo-controlled Clinical Trial of the Effect of Noni Juice on Lipid Peroxidation-derived DNA Adducts in Current Heavy Smokers
Brief Title: Effect of Noni Juice on Lipid Peroxidation-derived DNA Adducts in Heavy Smokers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tahitian Noni International, Inc. (Industry)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNI-UIC-01
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: DNA Damage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 59 mL noni juice (Experimental): Ingestion of 59 mL of Tahitian Noni® juice (mixture of noni juice and grape and blueberry juices) twice daily (118 mL daily total) for 30 days.
  Interventions: Dietary Supplement: Noni juice
- Placebo (Placebo Comparator): Ingestion of 59 mL of placebo (mixture of grape and blueberry juices and natural cheese flavor) twice daily (118 mL daily total) for 30 days.
  Interventions: Dietary Supplement: Placebo
- 29.5 mL noni dose (Experimental): Ingestion of 29.5 mL of Tahitian Noni® juice (mixture of noni juice and grape and blueberry juices) daily for 30 days.
  Interventions: Dietary Supplement: Noni juice

INTERVENTIONS:
Dietary Supplement: Noni juice — Ingestion of noni juice, a source of iridoids, daily for 30 days.
  Other Names: Tahitian Noni® Juice; Tahitian Noni® Original Bioactive; Thrive Adaptogenics Original
  Arms: 29.5 mL noni dose; 59 mL noni juice
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine if noni juice reduces lipid hydroperoxide (LOOH) and malondialdehyde (MDA) derived-DNA adducts, markers of oxidative DNA damage, in peripheral blood lymphocytes of cigarette smokers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years in age, smoker of more than 20 cigarettes per day, a smoking history exceeding one year, and willing to complete a one month trial.

Exclusion Criteria:

* concurrent use, or use in the previous three months, of prescription medication or antioxidant vitamins

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2000-09; Primary Completion 2005-11 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
LOOH and MDA-DNA adducts | 1 month
  LOOH and MDA-DNA adducts in lymphocytes immediately prior to intervention and at completion of intervention.

SECONDARY OUTCOMES:
adverse events | 1 month
  Adverse health events

CONTACTS AND LOCATIONS:
Overall Officials: Mian-ying Wang, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois College of Medicine at Rockford, Rockford, Illinois, United States